CLINICAL TRIAL: NCT06537128
Title: Internet-delivered Cognitive-Behavioral Therapy for Adolescents With Autism and Anxiety: Development and Evaluation of Learning to Understand and Navigate Anxiety-Adolescent
Brief Title: Internet-delivered Cognitive-Behavioral Therapy for Adolescents With Autism and Anxiety
Acronym: LUNA-A
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Eric A Storch, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-55617
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder; Autism; Anxiety; Anxiety Disorders; Generalized Anxiety Disorder; Social Anxiety Disorder
Keywords: Cognitive Behavioral Therapy; Adolescents; Autism; Anxiety
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Anxiety Disorders; Generalized Anxiety Disorder; Phobia, Social | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized assignment to one of two conditions
Who Masked: Outcomes Assessor
Masking Description: Independent evaluators will be blind to which group participants are randomized into.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LUNA-Adolescent (Active Comparator): Dyads in the Learning to Understand and Navigate Anxiety-Adolescent (LUNA-Adolescent) group will receive internet-based cognitive behavioral therapy (LUNA-Adolescent), which includes 12 weekly treatment modules, 6 bi-weekly, 30-minutes telehealth visits, and email check-ins.
  Interventions: Behavioral: LUNA-Adolescent
- Treatment as Usual (Placebo Comparator): Dyads in the standard-care cognitive behavioral therapy (CBT) group will receive 12 weekly sessions of transdiagnostic CBT for anxiety in autistic youth.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: LUNA-Adolescent — Learning to Understand and Navigate Anxiety-Adolescent (LUNA-Adolescent) includes parent-led, internet-based cognitive behavioral therapy (CBT) for anxiety among autistic youth.
  Other Names: Internet-based Cognitive Behavioral Therapy
  Arms: LUNA-Adolescent
Behavioral: Treatment as Usual — Treatment as Usual includes 12 weekly sessions of transdiagnostic cognitive behavioral therapy (CBT) for anxiety in autistic youth.
  Arms: Treatment as Usual

SUMMARY:
Anxiety is very common in autistic youth. Cognitive behavioral therapy (CBT) is the recommended treatment for both autistic and typically-developing (TD) youth with anxiety, yet most families cannot access CBT due to cost, practicalities of attending in-person treatment sessions, and a shortage of trained providers, especially in rural areas. The goal of this project is to increase access to care for families of autistic adolescents with anxiety through an internet-based treatment model.

DETAILED DESCRIPTION:
Autism affects 2-3% of youth, approximately half of whom experience a co-occurring anxiety disorder. Anxiety disorders in autistic youth are associated with significant life impairment and worsening trajectory without treatment. Cognitive behavioral therapy (CBT) is the recommended treatment for both autistic and typically-developing (TD) youth with anxiety, yet most families cannot access CBT due to cost, practicalities of attending in-person treatment sessions, and a shortage of trained providers, especially in rural areas. Access to CBT is particularly limited for Hispanic or Spanish-speaking families due to lack of services provided in Spanish. Internet-delivered therapies such as iCBT provide low intensity but effective intervention and overcomes barriers such as cost, travel, time from work/school, and stigma. Studies suggest that iCBT protocols for anxious typically-developing youth demonstrate moderate to strong effect sizes relative to control groups. However, until recently, such treatment models have not been developed with stakeholder engagement to be personalized for autistic children with anxiety and their families, including for those families that speak Spanish. In a previous Texas Higher Education Coordinating Board (THECB) funded work, a parent-led iCBT intervention for anxiety among autistic youth, Learning to Understand and Navigate Anxiety (LUNA) was developed. Over 60% of participants demonstrated response to treatment, yet children responded better than adolescents. Family feedback indicated that the materials were not developmentally appropriate for adolescents, necessitating further efforts to develop and evaluate an adapted version which is personalized to the unique needs of autistic adolescents with anxiety. The goal of this project is to increase access to care for families of autistic adolescents with anxiety through an internet-based treatment model (LUNA-Adolescent). This treatment model, developed by the study team, consists of an interactive website with both parent- and adolescent-facing treatment materials, supported by brief therapist contact (e.g. telehealth sessions), both in English and Spanish. Specifically, this project will evaluate the efficacy and cost effectiveness of LUNA-Adolescent compared to standard-care CBT for anxiety. Overall, this study will provide important information regarding the potential benefits of internet-based, parent-led interventions for autistic adolescents with anxiety and its two different delivery models.

ELIGIBILITY:
Inclusion Criteria:

1. The child is between the age of 11-17 years old at enrollment.
2. The child is diagnosed with autism using a validated assessment (e.g., Autism Diagnostic Observation Schedule-Second Edition (ADOS-2), Childhood Autism Rating Scale-Second Edition (CARS-2), etc.).
3. The child has current, clinically significant anxiety and/or OCD as indicated by a clinician-administered standardized assessment (e.g. Mini-International Neuropsychiatric Interview for Children and Adolescents (MINI-KID) and Pediatric Rating Anxiety Scale modified for autism (PARS-ASD)).
4. Anxiety disorder is the child's primary/co-primary psychiatric diagnosis, and if secondary psychopathology is present, it will not interfere with treatment.
5. One parent/guardian over the age of 18 is able and willing to participate in assessment and treatment (e.g. has sufficient English/Spanish fluency, the decisional capacity to participate, and can commit to treatment duration).
6. The child is able to communicate verbally.
7. Participants are located in Texas.
8. The participant has an IQ above 69, based on the Kaufman Brief Intelligence Test-Second Edition (KBIT-2), another valid test or clinician judgement (e.g., a previous assessment conducted, and report shared with study team)

Exclusion Criteria:

1. The child has a diagnosis of a lifetime psychotic disorder and/or conduct disorder.
2. The child has significant, current suicidal/homicidal ideation and/or self-injury requiring medical intervention.
3. The child has limited verbal communication abilities (e.g., no independent verbal communication),
4. The child is receiving concurrent psychotherapy (including certain forms of social skills training, or behavioral interventions that target anxiety such as applied behavioral analysis).
5. The child has initiated new antidepressant medication within 12-weeks of assessment (4-weeks for stimulants/benzodiazepines/antipsychotics) or during therapy.
6. The child has changed psychotropic medication dosage within 4-weeks of assessment (2-weeks for stimulants/benzodiazepines/antipsychotics) or during therapy.
7. The child requires a higher level than can be provided through the study (e.g., significant, current suicidal ideation)

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 139 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Pediatric Anxiety Rating Scale modified for ASD (PARS-ASD) | Baseline (before treatment), during treatment (on average 6 weeks), post-treatment (on average 12 weeks), 1 month follow up
  Clinician-rated child anxiety severity throughout the past week. Each item is scored on a 0 to 5 scale (higher scores correspond to greater severity), yielding a total between 0 and 35. This measure has been modified for autistic youth

SECONDARY OUTCOMES:
Clinical Global Impression-Improvement (CGI-I) | during treatment (on average 6 weeks), post-treatment (on average 12 weeks), 1 month follow up
  Clinician-rated child psychopathology severity rating. A single item is scored 0-6 (0= very much improved; 6= very much worse).
Screen for Child Anxiety Related Disorders (SCARED) | Baseline (before treatment), post-treatment (on average 12 weeks), 1 month follow up
  Parent and child self-report measure assessing anxiety symptoms including subscales for separation anxiety disorder, generalized anxiety disorder, social anxiety disorder, panic disorder or significant somatic symptoms, and significant school avoidance. A single item is scored on a 3 point Likert scale ranging from 0 (not true or hardly ever true) to 2 (very true or often true).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Storch, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No